CLINICAL TRIAL: NCT04699565
Title: Characterization of Patients With Post-ischemic Left Ventricular Dysfunction
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Paolo G Camici MD FACC, Prof Paolo G. Camici MD, FACC, IRCCS San Raffaele
Other Study IDs: VavirimS
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Left Ventricular Diastolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance — Evaluate the predictive value of myocardial viability measured with cardiac magnetic resonance for the identification of LV REM 6 months after STEMI

SUMMARY:
This is an observational, prospective, multicenter study (12 hospitals belonging to the Italian Cardiology Network) in patients with STEMI ST elevation myocardial infarction (STEMI) treated successfully with primary percutaneous coronary intervention (PCI), that will be followed for 12 month after the acute event, in order to ascertain the predictive value of myocardial viability measured with cardiac magnetic resonance (1.5 T; based on the transmural distribution of late enhancement in the infarcted segments) for the identification of left ventricular (LV) remodelling (REM) 6 months after STEMI.

DETAILED DESCRIPTION:
The present study is divided into 3 appointments following the standard inpatient stay for the index event (STEMI).

T0: Inpatient stay for index STEMI. Assessment of eligibility for participation in the study:

* STEMI diagnosis
* Primary PCI
* Confirmation at second-day transthoracic echocardiogram and pre-discharge echocardiogram of left ventricular dysfunction
* Biomarker assay

Visit 1 (V1): between 30 and 40 days post-STEMI. Clinical evaluation and performance of cardiac MRI with paramagnetic contrast agent (gadolinium) for measurement of infarct territory size and myocardial viability.

Visit 2 (V2): 6 months after STEMI. Clinical evaluation and second cardiac MRI, without contrast medium, for measurement of left ventricular volumes and consequently for measurement of the presence of adverse left ventricular remodeling.

Visit 3 (V3): 12 months after STEMI. Clinical re-evaluation with collection of data regarding events of interest for secondary endpoint. Performance of transthoracic echocardiogram.

The examinations and follow-up visits included in this study are part of clinical practice for treatment and risk assessment in patients who suffered STEMI with the exception of cardiac MRI without contrast medium at 6 months.

Cardiac magnetic resonance (CMR) data (1 month and 6 months) will be centrally analyzed post hoc at the MRI center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI (first episode) (defined according to European Society of Cardiology Guidelines 2017) with symptom onset within 12h (Class I), or >12h <48h (Class IIa), successfully treated by primary PCI.
* Patients with regional systolic dysfunction of 2 or more adjacent segments of the left ventricle, in the territory of the culprit artery, documented by echocardiogram on day 2 (Echo1) and confirmed at pre-discharge follow-up (Echo2).

Exclusion Criteria:

* Patients with documented prior myocardial infarction. In the event that cardiac MRI examination performed one month after STEMI shows areas of late enhancement even in segments of the left ventricle other than those subtended by the culprit artery, the patient will be allowed to continue the study if he or she does not have significant left ventricular dilatation and has no symptoms of heart failure;
* Patients with known cardiomyopathy;
* Patients with malignant neoplasia or systemic pathology with a "quoad vitam" prognosis of less than 1 year;
* Patients with known active infectious disease;
* Patients who are unable to express valid informed consent at the time of enrollment;
* Patients with specific contraindications to the performance of cardiac MRI, including:

Wearers of non-resonance-compatible devices; Previous surgery with placement of non-resonance-compatible vascular clips Claustrophobic patients; Patients with allergies and/or other specific contraindications to the use of paramagnetic contrast agents (gadolinium).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute ST-segment elevation myocardial infarction (STEMI) treated with effective primary angioplasty (PCI)
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Adverse left ventricular remodeling 6 month after index event | Six months
  Adverse LV remodeling, defined as ≥12% increase in enddiastolic LV volume 6 months after STEMI
  Diagnostic accuracy of CMR performed 1 month after STEMI to predict actual LV remodeling at 6 months

SECONDARY OUTCOMES:
Incidence of cardiovascular adverse event 1 year after STEMI in patients with evidence of left ventricular remodeling at 6 months compared with those without remodeling | Twelve months
  Incidence of the composite endpoint of death from cardiovascular causes, re-infarction, nonfatal stroke, new coronary revascularization interventions, development of heart failure, and new hospitalizations for cardiovascular causes 1 year after STEMI in patients with evidence of left ventricular remodeling at 6 months compared with those without remodeling.
Incidence of cardiovascular adverse events 1 year after STEMI in patients stratified with respect to total left ventricular viability | Twelve months
  Incidence of cardiovascular adverse events 1 year after STEMI in patients stratified with respect to total left ventricular viability (i.e., percent left ventricular volume free of late enhancement (the total volume of the left ventricle showing no enhancement minus the volume of left ventricular myocardium with evidence of late enhancement).
Predictivity of the presence of microvascular obstruction | Six months
  Predictivity of the presence of microvascular obstruction (MVO) in the infarcted area measured with CMR 1 month after STEMI on the development of LV remodeling at 6 months.
Predictivity of circulating biomarkers measured in the acute phase on the development of left ventricular remodeling six months after STEMI | Six months
  Predictivity of circulating biomarkers [NT-proBNP, troponin T (TnT), PCR], measured in the acute phase on the development of left ventricular remodeling six months after STEMI.
Predictivity of circulating biomarkers measured in the acute phase on cardiovascular adverse events 12 months after STEMI | Twelve months
  Predictivity of circulating biomarkers (NT-proBNP, TnT, PCR), measured in the acute phase on cardiovascular adverse events 12 months after STEMI.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Camici, MD, FACC, Principal Investigator — Ospedale San Raffaele
Locations (10):
- Italy (10):
  - IRCCS AOU San Martino, Genova
  - IRCCS Centro Cardiologico Monzino, Milan
  - IRCCS Fondazione Ca' Granda, Milan
  - IRCCS Istituto Auxologico Italiano, Milan
  - Paolo Camici, Milan
  - Irccs Sdn, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - IRCCS Fondazione Policlinico Gemelli, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Multimedica, Sesto San Giovanni

IPD SHARING:
Plan to Share IPD: No